CLINICAL TRIAL: NCT05614440
Title: The Effects of Tramadol Combined With Local Anesthesia on Pain After the Surgical Extraction of Third Molars
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 153-2011
Record Dates: First submitted 2022-10-31; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Pain After the Surgical Extraction of Third Molars
Keywords: tramadol; third molar extraction; analgesia
MeSH Terms: conditions — Agnosia | interventions — Anesthetics, Local; Tramadol; Carticaine

STUDY DESIGN:
Intervention Model Description: The patients were randomly divided into the following two groups using the sealed envelope method.
Who Masked: Care Provider, Investigator
Masking Description: The solutions were prepared prior to the procedure by an anesthetic nurse who was not involved in the study. Investigator was blind to the groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Only local anesthetic group (Active Comparator)
  Interventions: Drug: Only local anesthetic
- Tramadol group (Experimental)
  Interventions: Drug: Local anesthetic + tramadol hydrochloride

INTERVENTIONS:
Drug: Local anesthetic + tramadol hydrochloride — Using tramadol hydrochloride and articain HCL for inferior alveolar nerve block
  Other Names: Articaine
  Arms: Tramadol group
Drug: Only local anesthetic — Using articain HCL for inferior alveolar nerve block
  Arms: Only local anesthetic group

SUMMARY:
The purpose of this study was to assess the efficacy of local anesthetic and tramadol combinations in the prevention of pain after the surgical extraction of third molars.

DETAILED DESCRIPTION:
The surgical removal of impacted third molar teeth is a procedure that is frequently encountered in oral and maxillofacial surgery practices. Pain following these operations is one of the most important factors affecting patient satisfaction. Several pain-management strategies are available. An alternative approach to pain control is to maximize drug levels at the tissue injury site by administering drugs locally.

Tramadol is a centrally acting opioid that provides good analgesia. It reduces the transmission of pain impulses by inhibiting serotonin and norepinephrine re-uptake. In addition to the systemic analgesic effects, the local anesthetic effects of tramadol on the peripheral nerves have been presented in multiple clinical and laboratory studies.

The aim of this study is to test the clinical efficacy of local anesthetic and tramadol combinations during and after the surgical extraction of the lower third molars.

ELIGIBILITY:
Inclusion Criteria:

* Score of ASA I-II (American Society of Anesthesiologists Physical Status I or II)
* Patient weights were less than 60 kg

Exclusion Criteria:

* Subjects who had taken a sedative, tranquillizer, or analgesic medication within the last 24 h,
* Sensitive to tramadol,
* Patients who needed an extra dose of anesthetic solution during the surgery

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2013-11-01 (Actual); Study Completion 2014-01-01 (Actual)

PRIMARY OUTCOMES:
Change in pain | 48 hours
  Postoperative pain was assessed using a Visual Analogue Scale (VAS) ranging from the absence of pain (score 0) to the most severe pain imaginable. VAS values were taken from the patient during; post-op 10 minutes, hour 1, hour 2, hour 4, hour 6, hour 12, hour 24, hour 48.

SECONDARY OUTCOMES:
Change in mean blood pressure | 60 minutes
  Change in mean blood pressure assessed in baseline (after anesthetic injection), minute 10minute, minute 20, minute 30, minute 40, minute 50, minute 60.
Change in heart rate | 60 minutes
  Change in heart rate assessed in baseline (after anesthetic injection), minute 10minute, minute 20, minute 30, minute 40, minute 50, minute 60.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Deshpande AA, Hemavathy OR, Krishnan S, Ahmed R. Comparison of effect of intra socket ketamine and tramadol on postoperative pain after mandibular third molar surgery. Natl J Maxillofac Surg. 2022 Jan-Apr;13(1):95-98. doi: 10.4103/njms.NJMS_141_20. Epub 2022 Apr 20. PMID 35911818
- [Background] Vallecillo C, Vallecillo-Rivas M, Galvez R, Vallecillo-Capilla M, Olmedo-Gaya MV. ANALGESIC EFFICACY OF TRAMADOL/DEXKETOPROFEN VS IBUPROFEN AFTER IMPACTED LOWER THIRD MOLAR EXTRACTION: A RANDOMIZED CONTROLLED CLINICAL TRIAL. J Evid Based Dent Pract. 2021 Dec;21(4):101618. doi: 10.1016/j.jebdp.2021.101618. Epub 2021 Jul 28. PMID 34922724
- [Background] Iqbal AM, Shetty P. Effect of Submucosal Injection of Tramadol on Postoperative Pain After Third Molar Surgery. J Oral Maxillofac Surg. 2019 Sep;77(9):1752-1759. doi: 10.1016/j.joms.2019.03.029. Epub 2019 Mar 29. PMID 31026419
- [Derived] Afat IM, Gonul O, Satilmis T. Tramadol combined with local anesthesia for postoperative pain in third molar surgery. BMC Oral Health. 2025 Oct 14;25(1):1610. doi: 10.1186/s12903-025-07011-0. PMID 41088090